CLINICAL TRIAL: NCT05106920
Title: How we Apply Ultrasound-guided Neuromodulation in Lower Back Pain Sufferers
Brief Title: Frequency Parameter Used to Apply Ultrasound-guided Neuromodulation Percutaneous
Acronym: Parameters NMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Seville (Other)
Responsible Party: Principal Investigator, Blanca de la Cruz Torres, Principal Investigator, University of Seville
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMP-Frequency
Record Dates: First submitted 2021-10-23; First posted 2021-11-04 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NMP 3 Hz (Experimental): Participants received the percutaneous electrical stimulation intervention. Specifically, this consisted of the application of a square wave biphasic electrical current, with 3 Hz frequency and a 250µs pulse width, at the maximal tolerable intensity, to cause an tolerable muscle contraction. The application was 10 stimulations of 10 seconds, with 10 seconds at rest between stimulations. A trained physiotherapist performed the PNM intervention.
  Interventions: Other: NMP
- NMP 10 Hz (Experimental): Participants received the percutaneous electrical stimulation intervention. Specifically, this consisted of the application of a square wave biphasic electrical current, with 10 Hz frequency and a 250µs pulse width, at the maximal tolerable intensity, to cause an tolerable muscle contraction. The application was 10 stimulations of 10 seconds, with 10 seconds at rest between stimulations. A trained physiotherapist performed the PNM intervention.
  Interventions: Other: NMP

INTERVENTIONS:
Other: NMP — Participants received the percutaneous electrical stimulation intervention. Specifically, this consisted of the application of a square wave biphasic electrical current, to cause a tolerable muscle contraction. The application was 10 stimulations of 10 seconds, with 10 seconds at rest between stimulations. A trained physiotherapist performed the PNM intervention.

SUMMARY:
In the daily clinical practice, one of the most frequent reasons for consultation physiotherapists is low back pain (LBP). Regardless of the origin of the problem, the approach from physiotherapy contemplates the reduction of pain through different procedures, including neuromodulation.

In the field of Physiotherapy, ultrasound-guided Percutaneous Neuromodulation (PNM) is defined as the application through a needle with ultrasound guidance of an electrical current at low or medium frequency, seeking a sensitive and / or motor response of a peripheral nerve in some point of its trajectory, or of a muscle in a motor point, with a therapeutic objective. The objective of the study is to analyze that the effect of PNM on the sciatic nerve produces statistically significant changes in pain, joint range and functionality in patients with chronic LBP. Forty subjects will be recruited, which will be divided into 2 groups: group 1 to which PNM will be applied to the sciatic nerve at 250 microseconds, 3 Hz) during 90 seconds; group 2 to which PNM will be applied to the sciatic nerve in at 250 microseconds, 10 Hz during 90 second. The PNM intervention with NMP will consist in the single application of an asymmetric rectangular biphasic current.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Lower Back Pain
* Having no other therapy

Exclusion Criteria:

* Other pathology (discal hernia, injured limbs, neurological pathology)
* Belenophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Level of pain | From baseline measurement up to 1 week
  Measured by Visual Analogue Scale (0, no pain; 100, max pain)
Owestry questionnaire | From baseline measurement up to 1 week
  Lower back pain questionnaire. The final result is classified as minimal disability (0-20), moderate disability (21-40), severe disability (41-60), crippled (61-80) and bed-bound or exaggerating their symptoms (81-100).
Range of motion | From baseline measurement up to 1 week
  Measured by goniometer. Hip flexion, external and internal rotation range of motion
Y Balance Test | From baseline measurement up to 1 week
  Stability body
Strength | From baseline measurement up to 1 week
  Measured by dynamometer. Hip flexion, abduction, external and internal rotation muscle strength

CONTACTS AND LOCATIONS:
Locations (1):
- University of Seville, Seville, Spain